CLINICAL TRIAL: NCT02137915
Title: Long-Term Follow-up Study of the Phase I/II Safety and Preliminary Efficacy of Human Central Nervous System Stem Cells (HuCNS-SC) Subretinal Transplantation in Subjects With Geographic Atrophy of Age-Related Macular Degeneration
Brief Title: Long-Term Follow-up Safety Study of Human Central Nervous System Stem Cells in Subjects With Geographic Atrophy of Age-Related Macular Degeneration
Status: Terminated | Type: Observational
Why Stopped: Based on a business decision unrelated to any safety concerns.
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-N02-AMD
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Age-Related Macular Degeneration; Geographic Atrophy
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Human Central Nervous System Stem Cells
  Other Names: HuCNS-SC

SUMMARY:
This study is being done to determine the long-term safety and possible benefits of transplanted Human Central Nervous System Stem Cells (HuCNS-SC) for patients with Geographic Atrophy of Age-Related Macular Degeneration. This long-term follow-up study is limited to those individuals who received a transplant of HuCNS-SC cells into one of their eyes as part of the CL-N01-AMD study. No additional study product will be given in this 4-year long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed Study CL-N01-AMD
* Must be able to provide written informed consent prior to any study related procedures
* Agree to comply in good faith with all conditions of the study and to attend all required study visits

Exclusion Criteria:

* Inability to comply with study procedures or visits
* Since enrolling in Study CL-N01-AMD, have entered, or are about to enter another investigational study that, in the opinion of the Principal Investigator (PI), might confound study interpretation.
* Received off-study immunosuppressive agents in the lead-in study or are receiving any immunosuppressive agents since completing the lead-in study

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects with age-related macular degeneration (AMD) with GA who received transplantation of HuCNS-SC in Study CL-N01-AMD.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency and types of serious adverse events | At each of 11 visits over a period of 48 months

SECONDARY OUTCOMES:
Frequency and types of adverse events | At each of 11 visits over a period of 48 months

CONTACTS AND LOCATIONS:
Overall Officials: David Birch, Ph.D., Principal Investigator — Principal Investigator
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States